CLINICAL TRIAL: NCT04249492
Title: Multicentric Post-Market Clinical Follow-up (PMCF) Investigation to Determine Safety and Efficacy of a Hydrophobic EDOF Intraocular Lens (IOL) in Comparison to a Monofocal IOL
Brief Title: PMCF Study on EDOF (Isopure) vs Monofocal (Micropure) IOL
Acronym: PHY2001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Collaborators: targomedGmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHY2001
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cataract; Lens Opacities
Keywords: Intraocular Lens; EDOF; hydrophobic; IOL; monofocal
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind masking; Patient will not be informed which IOL model was implanted until end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL implantation experimental (Experimental): Experimental arm: Enhanced depth of focus (EDOF) intraocular lens.
  Interventions: Device: IOL implantation experimental (Isopure 1.2.3.)
- IOL implantation active comparator (Active Comparator): Comparator arm: Monofocal intraocular lens.
  Interventions: Device: IOL implantation active comparator (Micropure 1.2.3.)

INTERVENTIONS:
Device: IOL implantation experimental (Isopure 1.2.3.) — Implantation of trifocal IOL POD F GF consisting of light distribution order: far > intermediate > near
  Arms: IOL implantation experimental
Device: IOL implantation active comparator (Micropure 1.2.3.) — Implantation of trifocal IOL POD F GF consisting of light distribution order: far > near > intermediate
  Arms: IOL implantation active comparator

SUMMARY:
Multicenter, prospective, randomised, controlled, single-blind post-market clinical follow-up (PMCF) study to compare the clinical outcomes of an enhanced depth of focus (EDOF) IOL with the outcomes obtained with a monofocal lens. Implantation of the IOLs is bilaterally.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomised, controlled, single-blind post-market clinical follow-up (PMCF) study whereby patients undergoing routine cataract surgery will have bilateral implantation of Enhanced Depth of Focus intraocular lenses (Isopure 1.2.3.) or monofocal lenses (Micropure 1.2.3.). The patients will be randomized in a 1:1 ratio to receive the study or control lenses. Both IOLs, investigational device and control device, are CE approved and commercially available in the countries this clinical investigation is being carried out. The investigational device and all study products, including the devices used for the study examinations, will be used within the intended use specifications from the manufacturer. In addition, no invasive or other burdening examinations will occur for the patient.

The study will be carried out in up to five clinical centers in Europe and Asia.

The device under investigation (Isopure 1.2.3.) is a hydrophobic, glistening-free, acrylic EDOF intraocular lens (IOL) manufactured by the sponsor of this study, PhysIOL sa/nv. The control lens is the parent IOL, belonging to the same IOL family of this manufacturer. It is a hydrophobic, glistening-free, acrylic monofocal IOL (Micropure 1.2.3.). The IOLs will be implanted as part of the routine cataract surgery on patients suffering from cataract development.

Subjects participating in the trial will attend a total of maximum 11 study visits (1 preoperative, 1 or 2 operative and up to 8 postoperative) over a period of 12 months. If local requirements allow, preoperative and operative visit can be done on the same day. Subjects would have the option for unscheduled visits if required medically.

Primary endpoint data will be collected at the 120-180 days follow up visit. Secondary endpoint data will be collected at the 330-420 days follow up visit. Data interim analyses will be done after the last patient finished the 120-180 days postoperative examination to support the study publication plan.

ELIGIBILITY:
Inclusion Criteria:

* Cataractous eyes with no comorbidity;
* Calculated IOL power is within the range of the study IOLs;
* Male or female adults ages 45 years or older on the day of screening who have cataract(s) in one or both eyes;
* Regular corneal astigmatism ≤1.0 D (measured by an automatic keratometer)
* Clear intraocular media other than cataract;
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures;
* Signed informed consent.

Exclusion Criteria:

* Age of patient < 45 years;
* Regular corneal astigmatism >1.0 dioptres (measured by an automatic keratometer)
* Irregular astigmatism;
* Difficulty for cooperation (distance from their home, general health conditions);
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse;
* Subjects with AMD suspicious eyes as determined by OCT examination;
* Subjects who may be expected to require retinal laser treatment during the course of the study or at a greater risk of developing cystoid macular edema;
* Previous intraocular or corneal surgery;
* Traumatic cataract;
* History or presence of macular edema;
* Instability of keratometry or biometry measurements;
* Ocular hypertension or glaucoma;
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic / scotopic conditions);
* Expected complicated surgery;
* Significant dry eye.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
monocular Best Corrected Distance Visual Acuity (CDVA) under photopic light conditions on the first implanted eye. | 6 months (120-180 days) postoperative
  No statistically significant difference between the two study groups on monocular CDVA at 4-6 months follow up visit. A significance level of 0.05 or lower (p < 0.05) will be considered statistically significant. CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018.

SECONDARY OUTCOMES:
Manifested refraction | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2018. This data will also be used to calculate the manifested refractive spherical equivalent (MRSE)
Monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | Preoperative, 1 day (1-2 days) postoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  monocular UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Binocular UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Monocular CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Binocular CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Corrected Distance Visual Acuity (low contrast CDVA) using low contrast (10%) optotypes under photopic light conditions | 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Monocular CDVA using low contrast (10%) optotypes is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions. This test is performed using a low-contrast acuity chart with 10% contrast (using the Weber definition: [background - optotype]/background).
Monocular Uncorrected Intermediate Visual Acuity at 80cm (UIVA@80cm) under photopic light condition | 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Monocular UIVA@80cm is measured with ETDRS charts placed in 80cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Intermediate Visual Acuity at 80cm (UIVA@80cm) under photopic light condition | 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Binocular UIVA@80cm is measured with ETDRS charts placed in 80cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Intermediate Visual Acuity at 80cm (DCIVA@80cm) under photopic light conditions | 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Monocular DCIVA@80cm is measured with ETDRS charts placed in 80cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Distance Corrected Intermediate Visual Acuity at 80cm (DCIVA@80cm) under photopic light conditions | 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Binocular DCIVA@80cm is measured with ETDRS charts placed in 80cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Distance Visual Acuity at 80cm (low contrast DCIVA@80cm) using low contrast (10%) optotypes under photopic light conditions | 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Monocular DCIVA@80cm using low contrast (10%) optotypes is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions. This test is performed using a low-contrast acuity chart with 10% contrast (using the Weber definition: [background - optotype]/background).
Monocular Uncorrected Intermediate Visual Acuity at 66cm (UIVA@66cm) under photopic light condition | 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Monocular UIVA@66cm is measured with ETDRS charts placed in 66cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Intermediate Visual Acuity at 66cm (UIVA@66cm) under photopic light condition | 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Binocular UIVA@66cm is measured with ETDRS charts placed in 66cm distance. The examination is done without corrective glasses and according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Intermediate Visual Acuity at 66cm (DCIVA@66cm) under photopic light conditions | 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Monocular DCIVA@66cm is measured with ETDRS charts placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Distance Corrected Intermediate Visual Acuity at 66cm (DCIVA@66cm) under photopic light conditions | 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Binocular DCIVA@66cm is measured with ETDRS charts placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Distance Visual Acuity at 66cm (low contrast DCIVA@66cm) using low contrast (10%) optotypes under photopic light conditions | 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative
  Monocular DCIVA@80cm using low contrast (10%) optotypes is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions. This test is performed using a low-contrast acuity chart with 10% contrast (using the Weber definition: [background - optotype]/background).
Binocular Distance Corrected Near Visual Acuity at 40cm (DCNVA) under photopic light conditions | 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  Binocular DCNVA is measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Defocus Curve | 1 month (30-60 days) postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -2.5 D to +1.5 D in 0.5 D steps. In addition the following vergence values are measured: -0.25 D and +0.25 D. This examination is performed monocularly.
Binocular Defocus Curve | 6 months (120-180 days) postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -2.5 D to +1.5 D in 0.5 D steps. In addition the following vergence values are measured: -0.25 D and +0.25 D. This examination is performed binocularly.
Binocular Contrast Sensitivity under photopic light conditions | 6 months (120-180 days) postoperative
  Contrast Sensitivity under photopic light conditions using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions | 6 months (120-180 days) postoperative
  Contrast Sensitivity under mesopic light conditions using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions and using a glare source | 6 months (120-180 days) postoperative
  Contrast Sensitivity under mesopic light conditions with a glare source using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Halo and Glare Simulator | preoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  A Halo and Glare simulator software (Eyeland Design Network GmbH, Germany) will be used to assess the subjective perception of photic phenomena. The patients will be asked to adjust the halo and glare level in a simulated image to the amount they perceive such photic phenomena. This test is performed pre- and postoperatively. The preoperative outcomes deal as a baseline measurement.
Patient reported outcomes - Quality of Vision questionnaire [McAlinden et al, 2010] | preoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  To assess the subjective perception of disturbances by photic phenomena, the validated and verified Quality of Vision (QoV) questionnaire will be used.
  This questionnaire is a linear-scaled 30-item instrument and is designed with 10 symptoms rated in each of three scales (frequency, severity, and bothersome).
  The QoV Questionnaire provides a QoV score in terms of symptom frequency, severity, and bothersome [McAlinden et al, 2010].
Patient reported outcomes - Catquest-9SF 2011 questionnaire [Lundström et al, 2009] | preoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  To assess if difficulties in daily life occur due to impaired sight. This questionnaire is 9-item Rasch-scaled instrument to assess subjective perception of visual impairment after surgery [Lundström et al, 2009].
Patient reported outcomes - Patient-Reported Spectacle Independence Questionnaire (PRSIQ) [Morlock et al, 2017] | preoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The PRSIQ is a patient-reported measure assessing spectacle independence following cataract surgery. The analyses conducted provide evidence for the use of the PRSIQ total score as a measure of spectacle independence [Morlock et al, 2017].
Aberrometry | preoperative, 6 months (120-180 days) postoperative
  Aberrometry outcomes are measured with a standard aberrometer. The following values will be evaluated in this study: Spherical aberrations, high order aberrations, lens tilt.
Pupil Size under photopic light conditions | preoperative, 6 months (120-180 days) postoperative
  Photopic pupil diameters are measured with a precision of at least +/-0.5 mm. For the photopic pupil diameters, eye illumination should be identical to that used for photopic contrast sensitivity testing. It is required that pupil measurements be made with an infrared pupillometer / CCD camera. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 10 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Pupil Size under mesopic light conditions | preoperative, 6 months (120-180 days) postoperative
  Mesopic pupil diameters are measured with a precision of at least +/-0.5 mm. For the mesopic pupil diameters, eye illumination should be identical to that used for mesopic contrast sensitivity testing. It is required that pupil measurements be made with an infrared pupillometer / CCD camera. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 10 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus examination with dilated pupil | preoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus
Slitlamp examination - Corneal status | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal Status
Slitlamp examination - Signs of inflammation | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  * Signs of inflammation
  * Anterior chamber cells,
  * Anterior chamber flare,
  * Cystoid macular oedema,
  * Hypopyon, and
  * Endophthalmitis.
Slitlamp examination - Pupillary block | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Pupillary block.
Slitlamp examination - Retinal detachment | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Retinal detachment.
Slitlamp examination - Status of anterior and posterior capsule | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Status of anterior and posterior capsule.
Slitlamp examination - IOL decentration | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL decentration.
Slitlamp examination - IOL tilt | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL tilt.
Slitlamp examination - IOL discoloration | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL discoloration.
Slitlamp examination - IOL opacity | Preoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL opacity.

OTHER OUTCOMES:
Intraocular pressure (IOP) measurement | Preoperative, 1 day (1-2 days) postoperative, 1 week (7-14 days) postoperative, 1 month (30-60 days) postoperative, 6 months (120-180 days) postoperative, 12 months (330-420 days) postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Keratometry | Preoperative
  Keratometric measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
IOL power and target refraction | Operative (day of surgery)
  The parameter of the implanted IOL must be recorded as well as the target refraction given by the IOL calculator. This parameter is needed to calculate the accuracy of achieving the target refraction. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus OCT | Preoperative, 1 month (30-60 days) postoperative
  An OCT (optical coherence tomography) image will be taken at the preoperative visit to identify AMD suspicious eyes that need to be excluded from this study. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Kretz, MD, Principal Investigator — Augentagesklinik Rheine
Locations (12):
- Hanusch Krankenhaus, Vienna, Austria
- Gemini Eye Clinic, Zlín, Czechia
- Germany (4):
  - Augen-Zentrum-Nordwest, Ahaus
  - Universitäts-Augenklinik Heidelberg, Heidelberg
  - Smile Eyes Augen + Laserzentrum, Leipzig
  - Augentagesklinik Rheine, Rheine
- Ireland (2):
  - Institute of Eye Surgery - Clane, Kildare
  - Institute of Eye Surgery, Waterford
- Asian Eye Institute, Makati City, Philippines
- Spain (3):
  - Oftalvist Alicante, Alicante
  - Miranza IOA Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McAlinden C, Pesudovs K, Moore JE. The development of an instrument to measure quality of vision: the Quality of Vision (QoV) questionnaire. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5537-45. doi: 10.1167/iovs.10-5341. Epub 2010 May 26. PMID 20505205
- [Background] Morlock R, Wirth RJ, Tally SR, Garufis C, Heichel CWD. Patient-Reported Spectacle Independence Questionnaire (PRSIQ): Development and Validation. Am J Ophthalmol. 2017 Jun;178:101-114. doi: 10.1016/j.ajo.2017.03.018. Epub 2017 Mar 22. PMID 28341605
- [Background] Lundstrom M, Pesudovs K. Catquest-9SF patient outcomes questionnaire: nine-item short-form Rasch-scaled revision of the Catquest questionnaire. J Cataract Refract Surg. 2009 Mar;35(3):504-13. doi: 10.1016/j.jcrs.2008.11.038. PMID 19251145